CLINICAL TRIAL: NCT03719027
Title: Prevalence of Chronic Thromboembolic Pulmonary Hypertension After Acute Pulmonary Embolism. History of the Diagnosis. (Preva-CTEPH) Study
Brief Title: Prevalence of Chronic Thromboembolic Pulmonary Hypertension After Acute Pulmonary Embolism : (Preva-CTEPH)
Acronym: Preva-CTEPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K161203J; 2017-A02047-46 (Other: ANSM)
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension (CTEPH); Pulmonary Embolism
Keywords: Prevalence and incidence of CTEPH after pulmonary embolism; history of diagnosis
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Retrospective and prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental): Patients followed-up after the diagnosis of pulmonary embolism (PE) Patients who survived after a PE and who consent to participate to the prospective interventional phase of the PREVA-CTEPH study have dyspnea assessment, EKG, and echocardiography to investigate the diagnosis of CTEPH
  Interventions: Diagnostic Test: Study population

INTERVENTIONS:
Diagnostic Test: Study population — Dyspnea assessment (NYHA functional class) EKG Echocardiography

SUMMARY:
The prevalence of chronic thromboembolic pulmonary hypertension (CTEPH) after pulmonary embolism (PE) varies widely (0.4% to 8.8%) in the literature. This large variation could be due to the inclusion of patients with pre-existing CTEPH revealed on the occasion of a recurrence of PE. However, the absence of hemodynamic data when diagnosing PE does not allow to distinguish these patients. A prospective multicentric study involving 146 patients showed that the majority of patients with CTEPH during follow-up had a pulmonary hypertension unknown at the time of PE diagnosis. It is necessary to confirm these results in a broader study.

The aim of this study is to evaluate the cumulative incidence of CTEPH after a PE.

DETAILED DESCRIPTION:
The patients selected in this study are patients with an objectively confirmed PE and previously included since at least 12 months in one of the studies of the INNOVTE network.

Patients who are alive at the time of the selection for the PREVA-CTEPH study are contacted by phone or by mail for inclusion in the prospective interventional part of the PREVA-CTEPH study. Patients who consent to participate to this prospective interventional phase of the PREVA-CTEPH study have dyspnea assessment, EKG, and echocardiography to investigate the diagnosis of CTEPH. Patients with dyspnea (NYHA >1) and/or a high or intermediate echocardiographic probability of pulmonary hypertension (ESC criteria) have a V/Q lung scan, a right heart catheterization and a pulmonary angiography to objectively confirm the diagnosis of CTEPH according to the current ESC guidelines.

Retrospective phase: All clinical (dyspnea, signs of right ventricular insufficiency...), echocardiographic and imaging (pulmonary angiography, V/Q lung scan) relevant data after the diagnosis of index PE are retrieved from the clinical chart of each patients alive at the time of the selection for the PREVA-CTEPH study and/or with a diagnosis of CTEPH confirmed after the diagnosis of index PE and/or if the patient don't consent to participate to the prospective interventional phase.

For patients died between the inclusion in one of the studies of the INNOVTE network and the time of the selection for the PREVA-CTEPH study, the date and the cause of death are recorded. The same data of the retrospective phase are retrieved.

All cases of CTEPH are adjudicated by an independent committee. In this case, initial Imaging data (CT pulmonary angiography and echocardiography) performed at the time of index PE diagnosis are retrieved for searching previous sign of CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Pulmonary embolism objectively confirmed
* Treated during at least 3 months with curative anticoagulant
* Previously included since at least 1 year in one of the studies of the INNOVTE network
* affiliated to the national social security
* after written informed consent

Exclusion Criteria:

* Patients with an objectively confirmed CTEPH before the diagnosis of index PE
* Follow-up impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2003 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Cumulated incidence of CTEPH | 30-day +/- 15 days after inclusion visit
  Cumulated incidence rate of CTEPH after pulmonary embolism

SECONDARY OUTCOMES:
Cumulated incidence of CTEPH in patients without previous signs of CTEPH at the time of index PE diagnosis | 30-day +/- 15 days after inclusion visit
  Cumulated incidence rate of CTEPH in patients without previous signs of CTEPH at the time of index PE diagnosis
Cumulated incidence of CTEPH in patients with previous signs of CTEPH at the time of index PE diagnosis | 30-day +/- 15 days after inclusion visit
  Cumulated incidence rate of CTEPH in patients with previous signs of CTEPH at the time of index PE diagnosis
Risk factors of CTEPH | 30-day +/- 15 days after inclusion visit
  Hazard ratio of risk factors independently and significantly associated with the diagnosis of CTEPH after pulmonary embolism
Complications associated with right heart catheterization | 30-day +/- 15 days after inclusion visit
  Complication rate of right heart catheterization
Complications associated with pulmonary angiography | 30-day +/- 15 days after inclusion visit
  Complication rate of pulmonary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SANCHEZ, MD, PhD, Principal Investigator — Université Paris Descartes
Locations (4):
- France (4):
  - CHU Jean Minjoz, Besançon
  - La Cavale Blanche, Brest
  - Hôpital européen Georges-Pompidou, Paris
  - Hôpital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient level meta-analysis for cumulative incidence rate and risk factors of CTEPH after PE

REFERENCES:
- [Result] Guerin L, Couturaud F, Parent F, Revel MP, Gillaizeau F, Planquette B, Pontal D, Guegan M, Simonneau G, Meyer G, Sanchez O. Prevalence of chronic thromboembolic pulmonary hypertension after acute pulmonary embolism. Prevalence of CTEPH after pulmonary embolism. Thromb Haemost. 2014 Sep 2;112(3):598-605. doi: 10.1160/TH13-07-0538. Epub 2014 Jun 5. PMID 24898545
- [Result] Ende-Verhaar YM, Cannegieter SC, Vonk Noordegraaf A, Delcroix M, Pruszczyk P, Mairuhu AT, Huisman MV, Klok FA. Incidence of chronic thromboembolic pulmonary hypertension after acute pulmonary embolism: a contemporary view of the published literature. Eur Respir J. 2017 Feb 23;49(2):1601792. doi: 10.1183/13993003.01792-2016. Print 2017 Feb. PMID 28232411